CLINICAL TRIAL: NCT05412966
Title: A Feasibility Study of PEAR-002b, a Novel Prescription Digital Therapeutic to Support Unobserved Buprenorphine Initiation and Adherence in Opioid Use Disorder Outpatients
Brief Title: Feasibility Study of Novel Prescription Digital Therapeutic Supporting Unobserved Buprenorphine Initiation & Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pear Therapeutics, Inc. (Industry)
Collaborators: Kaiser Foundation Research Institute (Other); Whitman-Walker Institute, Inc. (Other Government); National Institute on Drug Abuse (NIDA) (NIH); Hassman Research Institute, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEAR-002-101; R44DA049493 (NIH)
Record Dates: First submitted 2022-05-19; First posted 2022-06-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Opioid Use Disorder
Keywords: digital therapeutic
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PEAR-002B / reSET-O (Experimental): Digital Therapeutic
  Interventions: Device: PEAR-002B; Device: reSET-O

INTERVENTIONS:
Device: PEAR-002B — PEAR-002B is a novel prescription digital therapeutic to support unobserved buprenorphine initiation and adherence in Opioid Use Disorder
Device: reSET-O — reSET-O is an FDA-authorized mobile application treatment for opioid use disorder.

SUMMARY:
The purpose of this study is to assess feasibility of an at-home digital therapy designed to support buprenorphine initiation and adherence.

DETAILED DESCRIPTION:
The purpose of this study is to develop and evaluate the acceptability of a novel feature for use with the prescription digital therapeutic reSET-O.

This feature aims to improve the quality of treatment for opioid use disorder (OUD) patients starting buprenorphine initiation at home by providing new digital content and withdrawal symptom assessment to support them during this process.

This study will evaluate the acceptability of this new feature and assess success of at-home buprenorphine initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study specific assessments being performed
2. Male or female ≥18 years of age, inclusive
3. English proficiency to meaningfully participate in consent process, assessment and intervention
4. Meets clinical sites criteria for buprenorphine initiation (e.g. current opioid use)
5. Currently receiving buprenorphine outpatient treatment for OUD (Part 1) or wishing to start buprenorphine treatment
6. Capable of using common software applications on an internet-enabled mobile device (smart phone or tablet)
7. Interested in testing or using PEAR-002b
8. No prior history of reSET-O use
9. Has not participated in any other investigational drug trials within the past 30 days (or within 5 half-lives of study drug, whichever is longer) of enrollment
10. Is considered appropriate for participation by their clinician

Exclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of OUD and on methadone or naltrexone pharmacotherapy
2. DSM-5 diagnosis of OUD and already on buprenorphine
3. Planning to move out of the geographic area within 2 months
4. Unable to use English to participate in the consent process, the interventions, or assessments
5. Inability to comply with study procedures, due to severe medical conditions or otherwise
6. Currently receiving inpatient treatment for OUD
7. Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
PEAR-002B User Satisfaction Surveys | Week 1
  Satisfaction survey questions will be rated on a 5-point Likert scale ranging from "not at all satisfied" to "very satisfied". Descriptive statistics will be calculated for quantitative and ordinal endpoints
PEAR-002B Qualitative User Experience Interviews | Week 1
  Qualitative user experience interviews will be coded and analyzed using grounded theory methodology to identify common themes
Buprenorphine Initiation Success | Week 1
  Buprenorphine initiation success will be measured as the proportion of participants attending the post-buprenorphine initiation visit
Medication Adherence Rates | From Week 1 to Week 4
  Buprenorphine adherence rates as measured by proportion of total urine samples testing positive for buprenorphine or norbuprenorphine

SECONDARY OUTCOMES:
PEAR-002B Engagement Data | From Baseline to Week 1
  PEAR-002B engagement rates as measured by participant use patterns data
reSET-O Qualitative User Experience Interviews | Week 4
  Qualitative user experience interviews will be coded and analyzed using grounded theory methodology to identify common themes
reSET-O User Satisfaction Surveys | Week 4
  Satisfaction survey questions will be rated on a 5-point Likert scale ranging from "not at all satisfied" to "very satisfied". Descriptive statistics will be calculated for quantitative and ordinal endpoints

OTHER OUTCOMES:
Abstinence From Illicit Opioids | From Baseline to Week4
  Abstinence from illicit opioid use as measured by urine immunoassay to detect the presence/absence of opioids.
Treatment Retention | From Baseline to Week 4
  Treatment retention measured as time to drop out (last face to face contact with a patient) and analyzed using the Kaplan Meier method
Device Wearing Time | From Baseline to Week 4
  Device wearing time as measured by EmbracePlus wearable device data
Physiological Biomarker Data | From Baseline to Week 4
  Physiological data (e.g., heart rate) as measured by EmbracePlus wearable device

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hassman, Study Director — Hassman Research Institute, LLC
Locations (1):
- Hassman Research Institute, LLC, Berlin, New Jersey, United States

REFERENCES:
- [Derived] Luderer H, Enman N, Gerwien R, Braun S, McStocker S, Xiong X, Koebele C, Cannon C, Glass J, Maricich Y. A Prescription Digital Therapeutic to Support Unsupervised Buprenorphine Initiation for Patients With Opioid Use Disorder: Protocol for a Proof-of-Concept Study. JMIR Res Protoc. 2023 Jan 20;12:e43122. doi: 10.2196/43122. PMID 36662568